CLINICAL TRIAL: NCT00180713
Title: Simvastatin as a Treatment for Pulmonary Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WILK10554
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Simvastatin; Statins
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Control (Placebo Comparator): Placebo tablet once daily
  Interventions: Drug: Placebo
- Arm 2: Experimental (Experimental): Simvastatin 40mg od for 1 month, then uptitrated to 80mg od for 11 months.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40mg od for 1 month, then 80mg od for 11 months
  Other Names: Zocor
  Arms: Arm 2: Experimental
Drug: Placebo — Placebo tablet once daily.
  Arms: Arm 1: Control

SUMMARY:
The purpose of the study is to investigate the safety and efficacy of adding simvastatin to the current conventional treatment regimen for the management of pulmonary hypertension.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a disease that is characterised by progressive narrowing of the blood vessels of the lungs. This results in a pressure load on the heart and heart failure.

The narrowing is in part due to constriction but mostly due to structural changes in affected vessels. The structural changes affect all cell components of the vessel wall (the endothelial lining, the muscle layer and fibrous tissue) and can lead to local clot formation. In addition there is evidence of inflammation of the vessels and what is known as oxidative stress. The disease may occur with no obvious cause, when it is known as idiopathic, but it can also be associated with a variety of other diseases, including congenital heart disease, collagen vascular disease and HIV infection.

Current approaches to the treatment of pulmonary hypertension are unsatisfactory as they do not prevent disease progression and do not directly or adequately address many of the processes detailed above. Alternative or additional treatments are therefore required and an attrative approach is to use a statin (a 3-hydroxy-3-methylglutaryl-coenzymeA, or HMG-CoA, reductase inhibitor). Statins are widely used for their ability to lower blood cholesterol but increasing evidence indicates that these drugs also have direct effects on cell components of the vessel wall - including inhibiting inflammation, clot formation and oxidative stress - that might be beneficial in pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic PAH or PAH related to collagen vascular disease
* Age 18 years or over
* Receiving conventional therapy with diuretics, digoxin, warfarin, sildenafil and bosentan. Stable for 1 month
* 6 minute walk distance between 150m and 450m
* Modified NYHA functional class II or III

Exclusion Criteria:

* PAH from a cause other than permitted by entry criteria
* Change in PAH treatment in past 4 weeks
* Patients requiring prostanoid therapy
* Patients already taking a statin
* Clinically significant disturbance of liver function - AST or ALT >3xULM; bilirubin >1.5xULM
* Contraindication for a magnetic resonance scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wilkins, MD FRCP, Principal Investigator — Imperial College London
Locations (3):
- Department of Internal Medicine II, Klinikstrasse 36 D-35392, Giessen, Germany
- United Kingdom (2):
  - Royal Brompton Hospital, Sydney Street, London
  - Hammersmith Hospital, Du Cane Road, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilkins MR, Ali O, Bradlow W, Wharton J, Taegtmeyer A, Rhodes CJ, Ghofrani HA, Howard L, Nihoyannopoulos P, Mohiaddin RH, Gibbs JS; Simvastatin Pulmonary Hypertension Trial (SiPHT) Study Group. Simvastatin as a treatment for pulmonary hypertension trial. Am J Respir Crit Care Med. 2010 May 15;181(10):1106-13. doi: 10.1164/rccm.2009111-699oc. PMID 20460548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Control | Arm 2: Experimental
Started | 23 | 19
Completed | 18 | 16
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Control | Arm 2: Experimental | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Continuous [Mean (Full Range); unit: years] | 49.1 [24 to 73] | 43.2 [19 to 67] | 46.2 [19 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 8 | 2 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21 | 11 | 32
  Black | 0 | 1 | 1
  Other | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Right Ventricular Mass From Baseline
Description: As measured by cardiac magnetic resonance (the study is powered to detect an 8.5g difference in RV mass between the two treatments, based on reproducibility measurements of RV mass in healthy volunteers and patients)
Time Frame: 6 months post study treatment
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Arm 1: Control | Arm 2: Experimental
Number analyzed (Participants) | 23 | 19
grams | 3.9 (13.9) | -5.2 (11.3)
Statistical Analysis 1: Comparison: Arm 1: Control vs Arm 2: Experimental; Test type: Superiority; p = 0.028, ANOVA

2. Secondary Outcome: Change in 6-minute Walk Distance
Description: Change in distance achieved in 6 minute walk test from baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | Arm 1: Control | Arm 2: Experimental
Number analyzed (Participants) | 23 | 19
metres | 1 (57) | 3.1 (34.5)
Statistical Analysis 1: Comparison: Arm 1: Control vs Arm 2: Experimental; Analysis was performed by intention to treat at 6 months and per protocol at 12 months. Missing variables were replaced with medians or means (for variables missing at baseline) or with expected variables calculated on the percentage change between baseline and 24 weeks observed for the group (placebo or statin) as a whole (a technique called imputation). Missing variables accounted for less than 5% of the data and there were no missing CMR data at baseline; Test type: Superiority; p = 0.86, ANOVA

3. Secondary Outcome: Change in LV Mass
Description: Change in LV mass from baseline based on cardiac MRI
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Arm 1: Control | Arm 2: Experimental
Number analyzed (Participants) | 23 | 19
grams | -1.3 (10.9) | 1.7 (12.3)
Statistical Analysis 1: Comparison: Arm 1: Control vs Arm 2: Experimental; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4, ANOVA

4. Secondary Outcome: Circulating Levels of BNP
Description: Change in NT-proBNP levels compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: fmol/ml
Arm/Group | Arm 1: Control | Arm 2: Experimental
Number analyzed (Participants) | 23 | 19
fmol/ml | 49 (224) | -75 (167)
Statistical Analysis 1: Comparison: Arm 1: Control vs Arm 2: Experimental; Test type: Superiority; p = 0.041, ANOVA

5. Secondary Outcome: Change in Quality of Life Score
Description: Change in quality of life score from baseline as measured by Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) scored from 1-25, with higher scores indicating worse quality of life, the investigator reported the score change.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: change of score
Arm/Group | Arm 1: Control | Arm 2: Experimental
Number analyzed (Participants) | 23 | 19
change of score | 0 (4.7) | -1.6 (4)
Statistical Analysis 1: Comparison: Arm 1: Control vs Arm 2: Experimental; Test type: Superiority; p = 0.26, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of consent until the final study visit after a year.
Arm/Group | Arm 1: Control | Arm 2: Experimental
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/19
Other Adverse Events (participants affected / at risk) | 0/23 | 2/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Control (N=23) | Arm 2: Experimental (N=19)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Control (N=23) | Arm 2: Experimental (N=19)
Elevated Creatinine Kinase (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Standard terms of model non-commercial agreement for UK clinical research apply.